CLINICAL TRIAL: NCT07385859
Title: Prosthetic Satisfaction, Body Image, and Activity-Participation After Unilateral Lower Limb Amputation: An ICF-Based Analysis
Brief Title: Prosthetic Satisfaction, Body Image, and ICF Outcomes After Amputation
Acronym: ICF
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, MİNE PEKESEN KURTÇA, Assistant Professor, Ondokuz Mayıs University
Other Study IDs: OMU2025/148
Record Dates: First submitted 2026-01-16; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Transtibial Amputation - Unilateral; Lower Limb Amputation Below Knee; Body Image; Activities of Daily Living; ICF; Participation
Keywords: body image; Lower Limb Amputation; Activities of Daily Living; Social Participation; ICF
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with Unilateral Lower Limb Amputation: This cohort consisted of adults with unilateral transtibial lower limb amputation who had been using a prosthesis for at least one year. Participants were able to ambulate independently with a prosthesis and had no significant neurological or musculoskeletal conditions affecting mobility. No experimental intervention was applied as part of the study. All participants underwent a single-session assessment including self-report questionnaires evaluating prosthetic satisfaction, body image, and activity and participation based on the International Classification of Functioning, Disability and Health (ICF) framework.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention was administered as part of this study. This was an observational, cross-sectional study in which participants received no experimental treatment, device, or behavioral intervention. Data were collected during a single assessment session using self-report questionnaires to evaluate prosthetic satisfaction, body image, and activity and participation based on the International Classification of Functioning, Disability and Health (ICF) framework.

SUMMARY:
Lower limb amputation affects not only physical mobility but also psychological well-being, body perception, and involvement in daily and social life. Although prosthetic use is essential for restoring mobility, rehabilitation outcomes may be influenced by multiple physical and psychosocial factors. Understanding the relationships between prosthetic satisfaction, body image, and activity and participation may contribute to improved rehabilitation planning after amputation.

This observational, cross-sectional study aims to investigate the relationships between prosthetic satisfaction, body image, and activity and participation outcomes in adults with unilateral lower limb amputation who use a prosthesis. The study includes adults with unilateral transtibial amputation who have been using a prosthesis for daily activities.

Participants complete standardized self-report questionnaires to assess prosthetic satisfaction using the Trinity Amputation and Prosthesis Experience Scales, body image perception using the Amputee Body Image Scale, and activity and participation based on the International Classification of Functioning, Disability and Health (ICF) framework.

Activity outcomes focus on the ability to perform daily physical tasks such as standing, walking, stair negotiation, and mobility on different surfaces. Participation outcomes focus on involvement in daily routines, social interactions, transportation, work, and leisure activities.

Statistical analyses are planned to examine the associations between prosthetic satisfaction, body image, and activity and participation outcomes, while considering demographic and prosthesis-related factors such as age and duration of prosthesis use.

DETAILED DESCRIPTION:
This observational, cross-sectional study is conducted within the framework of the International Classification of Functioning, Disability and Health (ICF) to explore psychosocial and functional aspects of rehabilitation after unilateral lower limb amputation. The study focuses on understanding how prosthetic-related and person-related factors jointly relate to activity performance and participation in daily life.

Participants are adults with unilateral transtibial amputation who have been using a prosthesis in daily life. The study adopts a biopsychosocial perspective, emphasizing that rehabilitation outcomes after amputation are not determined solely by physical capacity or prosthetic characteristics but also by psychological factors such as body image and subjective satisfaction with the prosthesis.

Prosthetic satisfaction is evaluated as a multidimensional construct reflecting comfort, functionality, and personal acceptance of the prosthesis, while body image is considered a key psychosocial factor influencing movement confidence, self-perception, and engagement in daily and social activities. Activity and participation are examined as distinct but related domains in accordance with the ICF conceptual model.

By examining the relationships between prosthetic satisfaction, body image, and ICF-based activity and participation outcomes, this study aims to contribute to a more comprehensive understanding of rehabilitation after lower limb amputation. The findings are expected to support patient-centered rehabilitation planning by highlighting psychosocial targets alongside prosthetic and functional considerations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 64 years
* Unilateral transtibial lower limb amputation
* Use of a prosthesis for at least one year
* Ability to ambulate independently with a prosthesis
* Ability to read and understand questionnaires
* Voluntary participation with written informed consent

Exclusion Criteria:

* Congenital limb deficiency
* Bilateral lower limb amputation
* Neurological disorders affecting mobility (e.g., stroke, Parkinson's disease)
* Severe musculoskeletal conditions influencing gait or balance
* Recent prosthetic replacement within the previous six months
* Severe residual limb pain or uncontrolled phantom limb pain
* Cognitive or psychiatric impairment that could interfere with questionnaire completion

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consisted of adults aged 18 to 64 years with unilateral transtibial lower limb amputation who had been using a prosthesis for at least one year. Participants were able to ambulate independently with a prosthesis and had no major neurological, musculoskeletal, cognitive, or psychiatric conditions affecting mobility or questionnaire completion. All participants were recruited from a single prosthetics and orthotics center and provided written informed consent prior to participation.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
ICF-Based Participation Score | Baseline
  Participation was assessed using an ICF-based participation questionnaire consisting of 9 items related to involvement in daily routines and social life, including indoor and outdoor mobility, use of public transportation, self-care, helping others, interpersonal interactions, employment, and leisure activities. Each item was scored on a 5-point scale ranging from 0 (no difficulty) to 4 (complete difficulty). Lower scores indicate better participation.
ICF-Based Activity Score | Baseline
  Activity was assessed using an ICF-based activity questionnaire consisting of 8 items related to daily physical activities, including changing body position, standing, walking short and long distances, walking on different surfaces, negotiating obstacles, stair ambulation, and driving. Each item was scored on a 5-point scale ranging from 0 (no difficulty) to 4 (complete difficulty). Lower scores indicate better activity performance.
Body Image (Amputee Body Image Scale, ABIS) | Baseline
  Body image perception is evaluated using the Amputee Body Image Scale (ABIS), a 20-item self-report questionnaire designed to assess body image disturbance in individuals with limb amputation. Each item is rated on a 5-point Likert scale. Total scores range from 20 to 100, with higher scores indicating greater body image disturbance.
Prosthetic Satisfaction (Trinity Amputation and Prosthesis Experience Scales, TAPES) - Description | Baseline
  Prosthetic satisfaction is assessed using the Trinity Amputation and Prosthesis Experience Scales (TAPES). The prosthetic satisfaction domain evaluates satisfaction with prosthesis aesthetics, weight, and functional performance. Items are scored on a Likert scale, with total scores ranging from 3 to 15, and higher scores indicating greater prosthetic satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mine PEKESEN KURTÇA P PEKESEN KURTÇA, PhD, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the small sample size and the sensitive nature of the clinical and psychosocial information collected. Data sharing was not included in the original informed consent.